CLINICAL TRIAL: NCT05947552
Title: Variability of Serum Ferritin in CKD Patients and How These Variables May Affect the Treatment Decisions With Iron
Brief Title: Serum Ferritin In CKD Patients Serum Ferritin
Acronym: Ferritin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Mahmoud Osman, Assiut Lecturer, Assiut University
Other Study IDs: Serum Ferritin in CKD patients
Record Dates: First submitted 2023-05-23; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic kidney disease Patients: Chronic kidney Disease Patients stage 3 to stage 5
  Interventions: Drug: Serum ferritin

INTERVENTIONS:
Drug: Serum ferritin — Serum ferritin in CKD patients

SUMMARY:
Variability of serum ferritin in CKD patients and how these variables may affect the treatment decisions with iron supplements

DETAILED DESCRIPTION:
Serum ferritin has a wide range Variability in CKD patients this makes the use of serum ferritin as an indicator of iron deficiency is limited and mostly CKD is secondary to inflammation so serum ferritin as ferritin is an acute phase reactants so it will be very high in CKD patients ,

ELIGIBILITY:
Inclusion Criteria:

* ALL CKD patients stage 3 to 5 not on dialysis

Exclusion Criteria:

* inflammatory chronic diseases IDA Autoimmune disorders Liver diseases Malignancy Infections

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: ALL CKD patients who are not dialysis Stage 3 to 5
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-07-08 (Estimated); Primary Completion 2025-01-11 (Estimated); Study Completion 2025-01-11 (Estimated)

PRIMARY OUTCOMES:
to assess the role of serum ferritin in CKD patients din in CKD patients and how these variability | Recurring
  affect treatment decisions with iron

CONTACTS AND LOCATIONS:
Overall Officials: Hawaid Ab Nafady, Professor, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No